CLINICAL TRIAL: NCT02117102
Title: Effect of Use of a New Technique for Pediatric Urine Collection on the Length of Stay in the Emergency Department: Prospective Randomized Controlled Trial
Brief Title: Effect of Use of a New Technique for Pediatric Urine Collection in ER
Acronym: BLST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jeju National University Hospital (Other)
Responsible Party: Principal Investigator, Kang Jeong Ho, Emergency department, Jeju National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BLSTJEJUNUH
Record Dates: First submitted 2014-04-14; First posted 2014-04-17 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Urinary Tract Infection; Unspecified Fever
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bladder and lumbar stimulation (Experimental): Apply bladder and lumbar stimulation
  Interventions: Other: Bladder and lumbar stimulation technic
- Control group (No Intervention): Ordinary pediatric urine collection bag

INTERVENTIONS:
Other: Bladder and lumbar stimulation technic
  Other Names: BLST
  Arms: bladder and lumbar stimulation

SUMMARY:
Urinary tract infection is most common serious bacterial infection in children who admit into the emergency department (ED). However the collection of urine from young children is time consuming process. So many children and their family guardian waste time until medical disposition established.

In 2013, Maria Luisa Herreros Fernandez etc have suggested a new urine collection technique for newborn, that bladder and lumbar stimulation technique is fast and safe.

The aim of this study is to determine clinical efficacy of bladder and lumbar stimulation technique (BLST) for pediatric patient in ED.

DETAILED DESCRIPTION:
Bladder and lumbar stimulation technic

Step 1

- Oral or IV hydration : Aprropriate to the weight of the children

Step 2 - Bladder stimulation : Gentle tapping in the suprapubic area at a frequency of 100 taps per minute for 30 sec

Step 3

- Lumbar stimulation : Lumbar paravertebral zone in the lower back with a light circular massage for 30 sec

Both stimulation manoeuvres are repeated until micturition starts and a midstream urine sample can be caught in a sterile collector

ELIGIBILITY:
Inclusion Criteria:

* Children have unspecific fever and requiring and urine test

Exclusion Criteria:

* Initial shock state
* History of congenial urinary tract abnormality
* Parents who have declined taking part in the research

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 170 (Estimated)
Dates: Start 2014-05; Primary Completion 2014-09 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Success rate of bladder and lumbar stimulation techninc | 10 min
  Success is defined as the collection of a sample within 10 min of starting the stimulation manoeuvres

SECONDARY OUTCOMES:
Urine collection time | 3 hour
  Urine collection time is defined as time from ordering urine analysis to collection of a urine sample

CONTACTS AND LOCATIONS:
Overall Officials: Sung wook Song, Study Chair — Emergency department of Jeju national university hospital
Locations (1):
- Jeju national university hospital, Jeju City, Jeju Special Governing Province, South Korea

REFERENCES:
- [Background] Herreros Fernandez ML, Gonzalez Merino N, Tagarro Garcia A, Perez Seoane B, de la Serna Martinez M, Contreras Abad MT, Garcia-Pose A. A new technique for fast and safe collection of urine in newborns. Arch Dis Child. 2013 Jan;98(1):27-9. doi: 10.1136/archdischild-2012-301872. Epub 2012 Nov 21. PMID 23172785